CLINICAL TRIAL: NCT01339728
Title: Far-infrared Ray Illuminates Area of CV12 Acupoint to Investigate the Correlation of Skin Temperature and Skin Blood Flow Between CV12 Acupoint and Palm Central Part of Right Hand
Brief Title: Far-infrared Ray Effect on CV12 Acupoint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Ching-Liang Hsieh, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: DMR99-IRB-176-1
Record Dates: First submitted 2011-04-14; First posted 2011-04-21 (Estimated); Last update posted 2011-04-21 (Estimated); Status verified 2011-04

CONDITIONS: Reaction of Far Infrared Ray; Reaction of Skin Temperature

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: far-infrared ray — The duration of far-infrared ray is 20 minutes.

SUMMARY:
The purpose of the present study was to investigate the effect of far-infrared ray at CV12 acupoints area on the skin temperature and skin blood flow of palm central area of right hand, and the correlation between them.

DETAILED DESCRIPTION:
The purpose of the present study was to investigate the effect of far-infrared ray at CV12 acupoints area (the center is CV12 acupoints and the diameter is 10 cm) on the skin temperature and skin blood flow of palm central area of right hand, and the correlation between them.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult volunteers, male or female, ages between 20 and 40 years
* Neurological and physical examination without abnormal functions
* Far-infrared ray illumination without allergic reaction and contra- indication
* The participants were explained the objective of the study, agreed to accept the test and signed a letter of consent

Exclusion Criteria:

* People less than 20 years of age or more than 40 years
* Women in pregnant or lactating
* People with mental or behavioral anomalies could not follow the researchers
* People suffered from serious diseases such as myocardial infarction , heart failure, serious arrhythmia, hypertension, diabetes, autoimmune disease, chronic obstructive pulmonary diseases, and kidney failure, liver cirrhosis and cancer
* People suffered from limb edema and serious skin diseases
* People did not sign a letter of consent

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2010-10; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
far-infrared ray on CV12 acupoint area may increase the skin temperature | Each period was 20 min in duration

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Liang Hsieh, professor, Study Chair — China Medical University Hospital
Locations (1):
- China Medical University Hospital, Taichung, Taiwan